CLINICAL TRIAL: NCT03869879
Title: Mobility Rehab: A Feedback System for Mobility Rehabilitation for Older Adults
Brief Title: Mobility Rehab, a Therapist-assisted System for Gait Rehabilitation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Oregon Health and Science University (Other)
Collaborators: NorthWest Rehabilitations Associates (Unknown); APDM (Unknown)
Responsible Party: Principal Investigator, Martina Mancini, Assistant Professor, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: eIRB 16282
Record Dates: First submitted 2019-02-20; First posted 2019-03-11 (Actual); Last update posted 2020-05-11 (Actual); Status verified 2020-05

CONDITIONS: Parkinson Disease; Stroke; Multiple Sclerosis; Gait Disorders, Neurologic; Gait Disorder, Sensorimotor; Gait, Unsteady; Gait Ataxia; Gait, Stumbling; Gait, Shuffling
Keywords: gait; balance; falls; mobility; feedback
MeSH Terms: conditions — Parkinson Disease; Stroke; Multiple Sclerosis; Gait Disorders, Neurologic; Gait Ataxia

STUDY DESIGN:
Intervention Model Description: Eligible participants are randomized into two groups. One group will receive standard physical therapy for their gait or balance issue while the other will receive visual feedback-aided physical therapy.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Directing physical therapist will assess eligibility, and randomize participants. Physical therapy aide will conduct baseline measures (questionnaires, ABC scale, and 2min walk). The four treating physical therapists are split into two groups: two therapists will provide traditional physical therapy, while the two other therapists will provide visual feedback-aided therapy for their participants. A second, blinded physical therapy aide will complete a follow-up assessment (ABC scale, 2min walk).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Feedback-assisted physical therapy (Active Comparator): During a visual feedback session, therapists will spend 30min per session using the Mobility Rehab system for gait training with patients. Therapists may select modality, overground walking and/or treadmill, tasks (dual task, head turns, etc. as above) as appropriate for each patient. They will additionally spend 15min on endurance, strength, and static and dynamic balance in functional tasks.
  Interventions: Other: Feedback-assisted physical therapy
- Traditional physical therapy (Placebo Comparator): During a regular session, patients with gait impairment will work on gait with the following tasks for 30min: weights on ankles, dual tasks, UE support, partial body weight support, speed challenges, obstacles, and head turning. Therapists may select modality, overground walking and/or treadmill, tasks (dual task, head turns, etc. as above) as appropriate for each patient. They will additionally spend 15min on endurance, strength, and static and dynamic balance in functional tasks.
  Interventions: Other: Traditional physical therapy

INTERVENTIONS:
Other: Feedback-assisted physical therapy — The system uses unobtrusive, wearable, inertial sensors with real-time algorithms to provide real-time feedback on: step time asymmetry, foot clearance, arm swing, trunk lateral range, and foot strike angle during gait.
  Arms: Feedback-assisted physical therapy
Other: Traditional physical therapy — Therapists will treat these patients with traditional therapeutic modalities and practices.
  Arms: Traditional physical therapy

SUMMARY:
Phase II of this study includes a pragmatic clinical trial which will take place at Northwest Rehabilitation Associates (NWRA) in Salem, OR to verify the efficacy of the system in a physical therapy clinic.

DETAILED DESCRIPTION:
This Phase II project is a collaboration among: 1) APDM, an innovative small business that has successfully commercialized several innovative products to quantify human movement; 2) the Balance Disorders Laboratory in the department of Neurology at Oregon Health & Science University (OHSU); and 3) NorthWest Rehabilitation Associates (NWRA), a nationally-recognized outpatient rehabilitation center that will test the effectiveness of Mobility Rehab for adults with mobility disturbances.

The objective of this Phase II application is to prepare the Mobility Rehab system for commercialization and demonstrate its efficacy for mobility training. Our hypothesis is that feedback-based rehabilitation will be more effective than standard rehabilitation for gait in older adults with gait disturbances. In this Phase II, we will use a pragmatic clinical trial to evaluate the effectiveness of Mobility Rehab on 300 patients with various types of gait disturbances in a physical therapy clinic. In addition to visual feedback, the system will be optimized in Phase II to also provide verbal feedback commands for patients during training.

ELIGIBILITY:
Inclusion Criteria:

* 60-89 years old
* gait disturbances requiring physical therapy

Exclusion Criteria:

* unable to follow instructions (up to the practitioner's judgement)

Ages: 60 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2019-07-24 (Actual); Primary Completion 2021-05-30 (Estimated); Study Completion 2021-05-30 (Estimated)

PRIMARY OUTCOMES:
Activities-Specific Balance Confidence (ABC) Scale | Collected at a participant's baseline visit and final study visit, after an average of one month
  This questionnaire measures an individual's perception of their own balance. Individuals use a scale ranging from 0% to 100% in rating the amount of confidence they have in their balance during 16 hypothetical daily-life activities. A score of 100% would represent one being fully confident in their balance during a specific task, while a score of 0% would represent one having no confidence at all in their balance. Total score ranges from 0 to 1600.

SECONDARY OUTCOMES:
Gait speed | Collected at a participant's baseline visit and final study visit, after an average of one month
  Gait speed is measured through two instrumented, two-minute walks. The first walk is performed at the individual's casual walking pace and the second is performed at a pace the individual considers to be faster than their casual pace.

CONTACTS AND LOCATIONS:
Overall Officials: Martina Mancini, PhD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Northwest Rehabilitation Associate, Salem, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes
At the conclusion of the study raw data of motor tasks will be available, within the bounds allowed by HIPAA and institutional privacy policies.
Supporting Information: Study Protocol, SAP
Time Frame: At the conclusion of the project.
Access Criteria: Email study PI for IPD access

REFERENCES:
- [Derived] Silva-Batista C, Harker G, Vitorio R, Studer M, Whetten B, Lapidus J, Carlson-Kuhta P, Pearson S, VanDerwalker J, Horak FB, El-Gohary M, Mancini M. Mobility Rehab visual feedback system for gait rehabilitation in older adults. J Neuroeng Rehabil. 2023 Oct 24;20(1):144. doi: 10.1186/s12984-023-01260-2. PMID 37875971
- [Derived] Vitorio R, El-Gohary M, Pearson S, Carlson-Kuhta P, Harker G, Horak FB, Lapidus J, Studer M, Mancini M. Effectiveness of the Mobility Rehab System for Mobility Training in Older Adults: A Pragmatic Clinical Trial. Front Neurol. 2021 Sep 6;12:680637. doi: 10.3389/fneur.2021.680637. eCollection 2021. PMID 34552549